CLINICAL TRIAL: NCT00001837
Title: Sonographic Evaluation of the Effects of Raloxifene on the Uterus and Ovaries in Premenopausal Patients at High Risk for Developing Breast Cancer
Brief Title: Effects of Raloxifene on the Uterus and Ovaries of Premenopausal Patients
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990013; 99-CC-0013
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-10

CONDITIONS: Breast Cancer; Breast Neoplasm
Keywords: Sonohysterography; Color Doppler Sonography; Endometrium; Gynecologic; Menstrual Cycle; Premenopause
MeSH Terms: conditions — Breast Neoplasms

SUMMARY:
This research study is designed to work in cooperation with another study being conducted by the National Cancer Institute. The National Cancer Institute (NCI) is studying the effects of a drug called raloxifene on premenopausal women believed to have a high risk of developing breast cancer (98-C-0123).

In this study, researchers are interested in learning about the effects of raloxifene on the uterus and ovaries of the women participating in the NCI study. To do this researchers plan to conduct ultrasounds on the patients enrolled in the NCI study. In addition researchers plan to take samples of the lining of the uterus in these patients (endometrial biopsy) if found to be necessary.

The purpose of this study is to determine the reproductive effects of raloxifene on women who have normal functioning ovaries by taking ultrasounds of the ovaries and lining of the uterus (endometrium).

DETAILED DESCRIPTION:
Raloxifene is a selective estrogen receptor-modulating agent that has been recently approved by the FDA for the treatment of osteoporosis in postmenopausal patients. A phase II trial evaluating the safety and efficacy of raloxifene in premenopausal patients at high risk for developing breast cancer has been recently approved by the IRB (98-C-0123). In this protocol, for assessment of the effects of raloxifene on the endometrium and ovaries, patients are scheduled to be studied with transvaginal sonography and hysterosonography, once during their menstrual cycle at periodic intervals. They are also scheduled to have endometrial biopsies as indicated. It is known that all SERMs (clomiphene, tamoxifen and in one small study raloxifene) raise the area under the curve of estradiol levels throughout the cycle in premenopausal women. Our study is designed to study the reproductive effects of raloxifene in these young women with competent ovaries using sonography of the ovaries and endometrium, and correlating it with steroid hormone levels which would be obtained under protocol 98-C-0123.

ELIGIBILITY:
Women must be enrolled in NCI Study 98-C-0123.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1998-11; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fisher B, Costantino JP, Wickerham DL, Redmond CK, Kavanah M, Cronin WM, Vogel V, Robidoux A, Dimitrov N, Atkins J, Daly M, Wieand S, Tan-Chiu E, Ford L, Wolmark N. Tamoxifen for prevention of breast cancer: report of the National Surgical Adjuvant Breast and Bowel Project P-1 Study. J Natl Cancer Inst. 1998 Sep 16;90(18):1371-88. doi: 10.1093/jnci/90.18.1371. PMID 9747868
- [Background] Rayter Z, Gazet JC, Shepherd J, Trott PA, Fisher C, Svensson WE, Ford HT, A'Hern R. Gynaecological cytology and pelvic ultrasonography in patients with breast cancer taking tamoxifen compared with controls. Eur J Surg Oncol. 1994 Apr;20(2):134-40. PMID 8181578
- [Background] Wolf DM, Jordan VC. Gynecologic complications associated with long-term adjuvant tamoxifen therapy for breast cancer. Gynecol Oncol. 1992 May;45(2):118-28. doi: 10.1016/0090-8258(92)90273-l. PMID 1592278